CLINICAL TRIAL: NCT06251843
Title: Co-designing Support Strategies for Parents to Encourage Early Engagement With Health Services During the First Year Following Their Child's Diagnosis of Sickle Cell Disorder
Brief Title: Support Strategies for Parents During the First Year Following Their Child's Diagnosis of Sickle Cell Disorder
Status: Not yet recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: British Academy (Unknown); Sickle Cell Society (Unknown); King's College Hospital NHS Trust (Other); Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: Support_SCD
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease, SCD, sickle cell anaemia
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parents of children with sickle cell disorder: Parents whose child has been diagnosed with sickle cell disorder in the last 36 months
- Health professionals: Health professionals involved in the care of children sickle cell disorder

SUMMARY:
Background: Sickle cell disorder (SCD), the commonest genetic (faulty gene inherited from both parents) condition in the UK, affects mainly underserved groups. Babies with SCD must start treatments soon after birth to prevent them becoming unwell. Stigma, fear and inequalities can make it difficult for parents to accept their child's diagnosis and access appropriate treatment and support.

Aim: Develop strategies to improve support for parents during their child's first year of life following a SCD diagnosis to encourage early engagement with health services.

Method: Comprises two stages: (i) Determine why parents choose to engage with support or not (ii) Use this information to co-design strategies to ensure greater accessibility of support for parents during their child's first year of life.

Patient and Public Involvement: We are working with Sickle Cell Society and parents of children with SCD. Dissemination: Findings will be shared with support groups, charities, health professionals and academics.

ELIGIBILITY:
Inclusion Criteria:

* Parents whose children have been diagnosed with SCD via screening in the last 36 months
* Health professionals involved in the care of children with sickle cell disorder

Exclusion Criteria:

* Parents whose inclusion may be contradicted on psychosocial grounds or who are unable to give informed consent.
* Health professionals who do not have experience of caring for children with sickle cell disorder.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parents whose children have been diagnosed with SCD via screening in the last 36 months Health professionals involved in the care of children with sickle cell disorder
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Support strategies for families with a child with SCD | June 2025
  Co-design strategies to ensure greater accessibility of support for parents during their child's first year of life following a SCD diagnosis

SECONDARY OUTCOMES:
Existing support | July 2024
  Description of support strategies accessed nationally by parents during the first year following their child's SCD diagnosis
Parental reasons for accessing support | July 2024
  Reasons why parents choose to access support or not
Support priorities | Sept 2025
  priorities for improving accessibility to support for parents during their child's first year of life following a SCD diagnosis for the co-design groups

IPD SHARING:
Plan to Share IPD: Undecided
To be decided